CLINICAL TRIAL: NCT03156452
Title: A Multicentre Randomised Trial of First Line Treatment Pathways for Newly Diagnosed Immune Thrombocytopenia: Standard Steroid Treatment Versus Combined Steroid and Mycophenolate
Brief Title: Newly Diagnosed Immune Thrombocytopenia Testing the Standard Steroid Treatment Against Combined Steroid & Mycophenolate
Acronym: FLIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON/2016/6004; 2017-001171-23 (EudraCT Number); PB-PG-0815-20016 (Other Grant/Funding Number: National Institute for Health Research (NIHR))
Record Dates: First submitted 2017-05-02; First posted 2017-05-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Mycophenolic Acid; Prednisolone; Steroids

STUDY DESIGN:
Intervention Model Description: A multicentre, open label randomised clinical trial of MMF with steroid as a first line treatment for patients with ITP against the standard care pathway involving steroids alone as first line treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid & Mycophenolate mofetil 1st line (Experimental): Mycophenolate mofetil: 1 gm bd Non-IMP Steroid: 1mg/kg od 4 days (maximum of 100mg), 40mg od 2 weeks, 20mg od 2 weeks, 10mg od 2 weeks, 5mg od 2 weeks then 5mg alternate days 2 weeks.
  Interventions: Drug: Mycophenolate Mofetil
- Prednisolone (Steroid) alone 1st line (Active Comparator): Non-IMP steroid: 1mg/kg od 4 days (maximum of 100mg), 40mg od 2 weeks, 20mg od 2 weeks, 10mg od 2 weeks, 5mg od 2 weeks then 5mg alternate days 2 weeks.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 500 mg and 250mg tablets for oral administration
  Arms: Steroid & Mycophenolate mofetil 1st line
Drug: Prednisolone — 5mg tablets for oral administration
  Other Names: Steroid
  Arms: Prednisolone (Steroid) alone 1st line

SUMMARY:
This is a study of two treatment pathways [Standard steroid treatment versus combined steroid and Mycophenolate (MMF)] for subjects with newly diagnosed Immune Thrombocytopenia (ITP). ITP is an illness that causes bruising and bleeding due to a low platelet count (blood cells essential for normal clotting). Patients are first given high dose steroids but most suffer side effects (e.g. difficulty sleeping, weight gain, moods swings, high blood pressure and diabetes). In addition, the majority of patients become ill again when the steroids are stopped - only about 20% stay well long term. ITP is relatively rare, non-cancerous in nature and the rare impact on survival of ITP have prevented it from being a priority for research funding, with first line treatment being unsatisfactory and unchallenged for decades. This underestimates the profound adverse impact an ITP diagnosis and its treatment has on individual patients, many of whom are young.

MMF is often used as the next stage treatment for ITP and it works well. However, it can take up to 2 months to work during which patients continue to be at risk of bleeding, bruising, fatigue and usually need more steroids which they find intolerable. They are required to come to hospital for weekly blood tests and for many this impacts on work. We want to find out whether it would benefit more patients if everyone takes MMF at diagnosis instead of current practice (waiting for the illness to come back). We plan to test this by comparing the current way we treat patients to a new way with patients given MMF right at the start of their treatment. 120 patients from 20 different hospitals will be asked to take part and half will be randomly chosen for the new pathway.

DETAILED DESCRIPTION:
This is a multicentre, randomised clinical trial of MMF with steroid as a first line treatment for participants with ITP against the standard care pathway involving steroids alone as first line treatment. This is not a blinded study, therefore patients and research team will know which treatment arm the participant will be randomised to.

There are no additional appointments or separate trial visits for this trial. Participants will be seen at their usual hospital appointments, which may take slightly longer than they do usually to gather all the information needed to carefully record information for the trial and to see how the participants are.

Participants will be screened and given up to one week of steroid prior to randomisation to enable sufficient time to read information, discuss and ask questions with informed consent in an appropriate setting.

Participants will then be randomised to one of either two treatment pathways below and be asked to complete quality of life questionnaires:

1. Steroid +MMF pathway: 1mg/kg once daily prednisolone 4 days (maximum of 100mg), 40mg once daily 2 weeks, 20mg once daily 2 weeks, 10mg once daily 2 weeks, 5mg once daily 2 weeks then 5mg alternate days 2 weeks then stop, (Dexamethasone 20mg or 40mg daily for 4 days is an alternative option to prednisolone if deemed clinically more appropriate for individual circumstances).

   For the duration of steroid, patients will get a PPI (proton pump inhibitors) or H2 antagonist to protect against gastric bleeding and appropriate bone protection.

   From randomisation (alongside steroid), MMF 500mg twice daily starting dose then increased to 750mg twice daily after 2 weeks if tolerated and 1g twice daily after another 2 weeks if tolerated (4 weeks after starting).

   After 6 months of MMF therapy, all patients who have remained in complete remission (platelet count> 100 x10 9/L) will reduce the dose by 250mg (one capsule) each month. The aim is to continue on the lowest dose that achieves a haemostatic (safe) platelet count (platelet 50-100 x10 9/L) and to ensure that patients who have gone into a spontaneous remission do not continue to take the drug indefinitely.
2. Steroid only group: 1mg/kg once daily prednisolone 4 days (maximum of 100mg), 40mg once daily 2 weeks, 20mg once daily 2 weeks, 10mg once daily 2 weeks, 5mg once daily 2 weeks then 5mg alternate days 2 weeks then stop (Dexamethasone 20mg or 40mg orally daily for 4 days is an alternative option to prednisolone if deemed clinically more appropriate for individual circumstances).

For the duration of steroid, patients will get a PPI (proton pump inhibitors) or H2 antagonist to protect against gastric bleeding and appropriate bone protection.

Patients will be seen at the following time points after randomisation:

2 months, 4 months, 6 months and 12 months when the following procedures will take place:

* Laboratory tests (safety bloods)
* Date of treatment failure (refractory or relapse AND need for second line therapy). [If treatment failure occurs, choice of second line treatment will be individualised according to patient's clinical circumstances. Further steroid will be given according to clinical need. Hospital monitoring of platelet levels is part of routine care for ITP patients and we will collect these details from the medical notes without requiring patients to come in for additional samples to be taken. These locally collected samples may be collected monthly (or less often) for patients believed to be in stable remission and weekly at lower or declining platelet levels. We expect this to allow us to calculate the time in remission and time in relapse with reasonable accuracy over the 12 month follow up period].
* Vital signs
* Blood sugar results
* Medication side effects (including infections)
* Dose and duration of steroids
* Need for rescue or other treatments (including second or third line). [Emergency and rescue treatments will be permitted throughout the study. These include platelet transfusions, tranexamic acid and intravenous immunoglobulin. These are known not to impact on the natural history of ITP and it is recognised that they may be important for patient safety. The use of 'rescue treatments' will be recorded on the CRF]
* Hospital attendances or admissions
* Days off work
* Patient questionnaires: Quality of life assessment
* Immunoglobulins rechecked at 6 months and 12 months

In addition at Screening and 2 months, participants will have the option to give an extra blood sample for the Bristol Biobank (ancillary translational basic science studies). There is an additional patient information sheet and consent form for this. Participants can consent to enter the trial, but decline to have bloods taken for bio banking.

In addition at 6 and 12 months, immunoglobulins will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Patients (males and females) >16 years old with a diagnosis of ITP, a pl count <30x109/L AND a clinical need for first line treatment.
* Patients have provided written informed consent

Exclusion Criteria:

* The exclusion criteria include pregnancy and breastfeeding
* Patients with HIV, Hepatitis B or C, or Common Variable immunodeficiency.
* Women of child bearing potential require a pregnancy test result within 7 days prior to randomisation (as per 7.1 below) to rule out unintended pregnancy
* Contraindications to MMF or steroid (see SPC, Appendix 2) including patients with hypersensitivity to mycophenolate mofetil, mycophenolic acid or to any of the excipients or active significant infection
* Patients not capable of giving informed consent (e.g. due to incapacity)
* Patients unwilling to follow contraceptive advice if allocated to MMF treatment arm.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to treatment failure. | 1 year
  To include patients who are refractory (platelet count <30x109/L in spite of 2 weeks treatment in the steroid arm or platelet count <30x109/L in spite of 2 months treatment in the steroid +MMF arm) or who initially respond but then relapse (defined clinically as platelet count <30x109/L and need for further therapy).

SECONDARY OUTCOMES:
Medication side effects, toxicity and other adverse events (including infection episodes) | Up to 12 months post randomisation
  Most participants experience side effects from the medication, data will be collected on treatment side effects and adverse events as assessed by CTCAE V4.0
Bleeding events | up to 12 months post randomisation
  To be analysed as number of bleeding events per patient recorded by 12 months. In addition we will collect site and type of bleeding, treatment required for bleeding, whether hospital admission was required, whether ITP rescue treatments were needed to be used in the calculating of costs for the economic evaluation.
Remission rates | Up to 12 months post randomisation
  Platelet count >30 x109/L and at least 2 fold increase from baseline. Complete >100x10 9/L, partial 30-100x10 9/L
Time to relapse and time to next therapy | Up to 12 months post randomisation
  period of time between relapse and time of next therapy
Cumulative cortiocosteroid dose | Up to 12 months post randomisation
  Total steroid dose from randomisation
Need for rescue therapies | up to 12 months post randomisation
  To be analysed as number patients who required rescue therapies between randomisation and 12 months post randomisation. We will also record the mean number of rescue therapies, why they were needed their type and cost for use in the economic evaluation.
Need for splenectomy | Up to 12 months post randomisation
  Whether a participant has undergone splenectomy procedure
Socioeconomic costs | Up to 12 months post randomisation
  NHS, personal and social costs
Patient reported outcomes - Quality of Life | Up to 12 months post randomisation
  To be assessed using the utility score of the ICECAP (A) to calculate area under the curve using the trapezium method over a 12 month time frame from date of randomisation.
Patient reported outcomes - Fatigue | Up to 12 months post randomisation
  To be assessed using the utility score of the FACIT-F (Version 4) to calculate area under the curve over a 12 month time frame from date of randomisation.
Patient reported outcomes - Impact of bleeding | Up to 12 months post randomisation
  To be assessed using the utility score of the FACT-Th6 (Version 4) to calculate area under the curve over a 12 month time frame from date of randomisation.
Patient reported outcomes - Care Costs | Up to 12 months post randomisation
  To be assessed using the utility score of the Thrombocytopenia care costs V1 questionnaire to calculate area under the curve over a 12 month time frame from date of randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bradbury, Study Director — University of Bristol
Locations (1):
- University Hospital Bristol NHS Foundation Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stimpson ML, Wolf J, Charbit B, Williams EL, Lait PJP, Schewitz-Bowers LP, Lee RWJ, Bradbury CA. Systemic immunosuppression depletes peripheral blood regulatory B cells in patients with immune thrombocytopenia. Br J Haematol. 2024 Feb;204(2):644-648. doi: 10.1111/bjh.19144. Epub 2023 Oct 12. PMID 37823469
- [Derived] Bradbury CA, Pell J, Hill Q, Bagot C, Cooper N, Ingram J, Breheny K, Kandiyali R, Rayment R, Evans G, Talks K, Thomas I, Greenwood R. Mycophenolate Mofetil for First-Line Treatment of Immune Thrombocytopenia. N Engl J Med. 2021 Sep 2;385(10):885-895. doi: 10.1056/NEJMoa2100596. PMID 34469646
- [Derived] Pell J, Greenwood R, Ingram J, Wale K, Thomas I, Kandiyali R, Mumford A, Dick A, Bagot C, Cooper N, Hill Q, Bradbury CA. Trial protocol: a multicentre randomised trial of first-line treatment pathways for newly diagnosed immune thrombocytopenia: standard steroid treatment versus combined steroid and mycophenolate. The FLIGHT trial. BMJ Open. 2018 Oct 18;8(10):e024427. doi: 10.1136/bmjopen-2018-024427. PMID 30341143